CLINICAL TRIAL: NCT05276570
Title: A Phase 1/2a Study Evaluating the Effects of ARO-RAGE Inhalation Solution in Healthy Subjects and Patients With Inflammatory Lung Disease
Brief Title: Study of ARO-RAGE in Healthy Subjects and Patients With Inflammatory Lung Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ARORAGE-1001
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-RAGE (Experimental): ARO-RAGE Inhalation
  Interventions: Drug: ARO-RAGE
- Placebo (Placebo Comparator): (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-RAGE — single or multiple doses of ARO-RAGE by inhalation of nebulized solution
  Arms: ARO-RAGE
Drug: Placebo — calculated volume to match active treatment by inhalation of nebulized solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ARO-RAGE in normal healthy volunteers (NHVs) and in participants with inflammatory lung disease (asthma). In Part 1 of the study, NHVs will receive a single dose of ARO-RAGE or placebo. In Part 2 of the study, adult participants with asthma will receive 2 doses of ARO-RAGE or placebo. Additional NHVs may be randomized to receive 1 or 2 doses of ARO-RAGE or placebo at Sponsor discretion. Dose levels in Part 2 will be determined based on cumulative safety and pharmacodynamic data from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Normal pulmonary function tests at Screening (NHVs only)
* Confirmed diagnosis of asthma based on source verifiable medical record (asthma patients only)
* No abnormal finding of clinical relevance at Screening (other than asthma for asthma patients)
* Stable dose of asthma controller medications prior to Screening (asthma patients only)
* If on allergen-specific immunotherapy, participants must be on a stable maintenance dose
* Non-smoking
* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception. Males must not donate sperm during the study and for at least 12 weeks following the last dose of study drug
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Acute lower respiratory infection or asthma exacerbation within 30 days prior to first dose
* Positive COVID-19 test during Screening window
* Use of immunosuppressive medication within 90 days prior to first dose
* Receipt of any intranasal vaccine within 30 days prior to first dose
* Use of systemic corticosteroid therapy within 90 days prior to first dose
* Clinically significant health concerns (other than asthma in asthma patients)
* Human Immunodeficiency virus (HIV) infection, seropositive for Hepatitis B Virus (HBV), seropositive for Hepatitis C Virus (HCV)
* Uncontrolled hypertension
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study
* Use of illicit drugs
* Use of an investigational agent or device within 30 days prior to first dose

Note: additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug through the end of study (EOS; up to 113 days)

SECONDARY OUTCOMES:
Change from Baseline Over Time in Forced Expiratory Volume (FEV1) | Baseline through EOS (up to 113 days) or until serum soluble receptor for advance glycation end products (sRAGE) is ≥ 70% of baseline value
Change from Baseline Over Time in Forced Vital Capacity (FVC) | Baseline through EOS (up to 113 days) or until serum sRAGE is ≥ 70% of baseline value
Change from Baseline Over Time in Diffusing Capacity for Carbon Monoxide (DLCO) | Baseline through EOS (up to 113 days) or until serum sRAGE is ≥ 70% of baseline value
PK of ARO-RAGE: Maximum Observed Plasma Concentration (Cmax) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Time to Maximum Observed Plasma Concentration (Tmax) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to 24 Hours (AUC0-24) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to the Last Quantifiable Plasma Concentration (AUClast) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to Infinity (AUCinf) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Terminal Elimination Half-Life (t1/2) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Apparent Systemic Clearance (CL/F) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Apparent Terminal-Phase Volume of Distribution (VZ/F) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma
PK of ARO-RAGE: Recovery of Unchanged Drug in Urine Over 0 to 24 Hours (Amount Excreted; Ae) | Through 24 hours post-dose
PK of ARO-RAGE: Percentage of Administrated Drug Recovered in Urine Over 0 to 24 hours | Through 24 hours post-dose
PK of ARO-RAGE: Renal Clearance (CLr) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs, and up to 24 hours post-dose for participants with asthma

CONTACTS AND LOCATIONS:
Locations (8):
- Research Site 1, Nedlands, Washington, Australia
- New Zealand (3):
  - Research Site 1, Auckland
  - Research Site 2, Auckland
  - Research Site 3, Auckland
- Poland (2):
  - Research Site 2, Krakow
  - Research Site 3, Oświęcim
- Research Site 1, Barcelona, Spain
- Research Site 1, Bangkok Noi, Bangkok, Thailand